CLINICAL TRIAL: NCT06118294
Title: Efficacy of Probiotics for Parkinson Disease (PD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has retired
Sponsor: Changhua Christian Hospital (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sheylin Wu, Principal Investigator, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 230723
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease (PD); Movement Disorders; Depression; Anxiety
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Depression; Anxiety Disorders | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: 300 Participants are assigned to the probiotics and a placebo group, under the double-blind trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): daily ingestion of 2 capsules of probiotics (>30 billion CFU/capsule)
  Interventions: Dietary Supplement: probiotics
- Placebo (Placebo Comparator): daily ingestion of 2 capsules which only contained 425 ± 25 mg microcrystalline cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: probiotics — >30 billion CFU/capsule
  Arms: Probiotics
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In previous clinical studies, PS128 has been reported to ameliorate motor deficits in Parkinson's disease (PD). PS23 has been reported to delay some age-related disorders.

On the basis of previous animal and clinical studies which hope that this study can support the theory of the gut-brain axis, and have the opportunity to realize the relationship between peripheral inflammation and neurodegeneration.

DETAILED DESCRIPTION:
The gut microbiota plays important roles in gastrointestinal homeostasis, essential physiological processes and CNS function, and affects the gut-brain axis via neural, immune and endocrine pathways giving rise to the microbiota-gut-brain-axis (MGBA). Combining the MGBA concept and the theory that Parkinson's disease (PD) is derived in the gut, researchers have studied the relationship between the gut microbiota and the PD neurodegenerative process. Probiotics are live microorganisms that confer health benefits on the host and can improve host physical and mental health by affecting MGBA homeostasis. Lactobacillus plantarum PS128 (PS128) and Lactobacillus paracasei PS23 (PS23) are specific probiotics, known as a psychobiotic, which has been demonstrated to alleviate depression- and anxiety-like behaviors in mouse model. Furthermore, PS128 alleviated motor deficits, nigrostriatal dopaminergic neuronal cell death, and striatal dopamine reduction in the MPTP mouse model of Parkinson's disease. In previous clinical studies, PS128 has been reported to ameliorate motor deficits in PD. PS23 has been reported to delay some age-related disorders.

On the basis of previous animal and clinical studies which hope that this study can support the theory of the gut-brain axis, and have the opportunity to realize the relationship between peripheral inflammation and neurodegeneration.

The eligible participants will be administered with probiotics capsules for 12 weeks. Symptoms of PD will be clinically evaluated before and after the treatment. Blood and stool samples will be collected before and after the intervention for biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* The age between 41-80 years old and at least the elementary education level.
* Diagnosed as a patient with Parkinson's disease of modified Hoehn and Yahr Stage between 1 and 3 as rated.

Exclusion Criteria:

* Diagnosed before 40 years old.
* Used probiotic products in powder, capsule, or tablet form within four weeks.
* Have taken antibiotics within four weeks.
* Those who are not suitable to participate in the research are judged by PI.

Ages: 41 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-08 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
UPDRS III | From Baseline to 12 Weeks Assessed
  The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients.
  The PART III is Motor sections.

SECONDARY OUTCOMES:
Clinical Global Impression scales of Severity rated by clinician（CGI） | From Baseline to 12 Weeks Assessed
  The CGIC is a single-item questionnaire that asks the investigator to assess a patient's PD symptoms at specific visits after initiating therapy. The CGIC uses a 7 point Likert Scale, ranging from very much worse (-3) to very much improved (+3), to assess overall response to therapy. A treatment success was defined as "much improved" or "very much improved" at the week 12 visit.
UPDRS I-IV | From Baseline to 12 Weeks Assessed
  The UPDRS scale refers to Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients.Scale UPDRS the sum of parts I, II and III ranges from 0 to 176. The UPDRS score has three components, each consisting of questions with 0-4 point scale. Part I assesses mentation, behavior, and mood; Part II assesses activities of daily; and Part III assesses motor abilities. Where 0 represents the absence of impairment and 4 represents the highest degree of impairment.
Q-LES-Q | From Baseline to 12 Weeks Assessed
  Participants who receive app-CBT will have greater improvement on quality of life, assessed using The Quality of Life, Enjoyment, and Satisfaction Questionnaire - Short Form (Q-LES-Q). The Q-LES-Q-SF is a self-report measure of subjective quality of life, containing Likert items ranging from 1 (Very Poor) to 5 (Very Good). Total scores are presented as a percentage of the maximum value (i.e., ranging from 0 to 100, with higher scores indicating greater quality of life).
Visual Analogue Scale for GI symptoms, VAS-GI | From Baseline to 12 Weeks Assessed
  Visual Analogue Scale for GI symptoms, VAS-GI (visual analogue scale, VAS 0-10) was designed to measure the response of symptoms and well-being in patients after taking probiotics
PGI-C | From Baseline to 12 Weeks Assessed
  The PGIC is a scale participants use to rate the level of change they have experienced following treatment. The PGIC is a 7-point scale from 1 (very much better) to 7 (very much worse).
PHQ-9 | From Baseline to 12 Weeks Assessed
  Measure for Major Depressive Disorder from questionnaire responses, to measure the prevalence of clinically significant depression defined as a PHQ-9 score of equal to or greater than 10.
Differences in the State and Trait Anxiety Index (STAI) | From Baseline to 12 Weeks Assessed
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Difference in Oxidative stress - blood level of HSCRP | From Baseline to 12 Weeks Assessed
  To assess inflammation indicators, used commercial kit human CRP (Cayman, Mich, USA) and Elisa reader (PerkinElmer, Massachusetts, USA) for analysis
Gut microbiota | From Baseline to 12 Weeks Assessed
  Collect the DNA of fecal flora to test the diversity and abundance of gut microbiota in Stool samples before and after probiotics
Level of Growth Differentiation Factor-15 | From Baseline to 12 Weeks Assessed
  Level of Growth Differentiation Factor-15
brain-derived neurotropic factor (BDNF) | From Baseline to 12 Weeks Assessed
  Measurement BDNF level in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital (CCH), Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided